CLINICAL TRIAL: NCT02930525
Title: Effect of High Flow Nasal Cannula vs. Standard Care on Respiratory Stability in Pediatric Procedural Sedation: A Randomized Controlled Pilot Trial
Brief Title: Effect of High Flow Nasal Cannula vs. Standard Care on Respiratory Stability in Pediatric Procedural Sedation
Acronym: HiFiPPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Freiburg (Other)
Responsible Party: Principal Investigator, Daniel Klotz, M.D., University of Freiburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 143/16
Record Dates: First submitted 2016-10-09; First posted 2016-10-12 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Respiratory Insufficiency
Keywords: apnea; children; hypercarbia; procedural sedation; HFNC
MeSH Terms: conditions — Respiratory Insufficiency; Apnea; Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (Active Comparator): Standard respiratory care. Oxygen delivered via low flow nasal cannula, increase of fractions of inspired oxygen to maintain desired oxygenation as defined per protocol.
  Interventions: Other: Standard respiratory care
- High Flow nasal cannula (Experimental): Application of humidified heated ambient air with flow rates adapted to body weight of respective subject. Incremental increase of fraction of inspired oxygen as appropriate to maintain oxygenation (defined as transcutaneous pulse oximetry above 93%).
  Interventions: Other: High Flow nasal cannula

INTERVENTIONS:
Other: High Flow nasal cannula — Application of humidified heated ambient air with flow rates adapted to body weight of respective subject. Incremental increase of fraction of inspired oxygen as appropriate to maintain oxygenation (defined as transcutaneous pulse oximetry above 93%).
  Arms: High Flow nasal cannula
Other: Standard respiratory care — Standard respiratory care. Oxygen delivered via low flow nasal cannula, increase of fractions of inspired oxygen to maintain desired oxygenation as defined per protocol.
  Arms: Standard care

SUMMARY:
Procedural sedation is an established and safe intervention and is widely used in diagnostic and therapeutic procedures for pediatric patients. Nonetheless, problems of the respiratory system such as upper airway obstruction, hypoventilation and apnea are frequent adverse events. We postulate that respiratory instability is less frequent in patients high flow nasal cannula vs. standard care on respiratory stability, i.e. low flow nasal cannula, in pediatric procedural sedation. The purpose of this pilot study is to estimate the effect of HFNC (high flow nasal cannula) on the respiratory instability in children undergoing upper gastrointestinal endoscopy under pediatric procedural sedation (PPS).

ELIGIBILITY:
Inclusion Criteria:

1. Age 6 years - 18 years
2. Undergoing pediatric non-emergency upper gastrointestinal endoscopy under sedation
3. Informed consent/assent for enrollment by parents/legal guardians/patient

Exclusion Criteria:

1. Congenital or acquired malformations involving the airways
2. Patients with the history of spontaneous pneumothorax or connectives tissue diseases (Marfan syndrome, Ehlers-Danlos-Syndrome)
3. Patients with a history of traumatic/iatrogenic air leak within the last 3 months before enrollment

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
Respiratory instability | Time frame from first applications of intravenous sedatives until finishing the intended procedure
  Number of episodes longer than 15 seconds with SpO2 < 93% and/ or pCO2 > 45 mmHg and/ or apnea (defined as cessation of airflow for > 15 seconds)

SECONDARY OUTCOMES:
Duration of respiratory instability | Time frame from first applications of intravenous sedatives until finishing the intended procedure
  Total duration of episodes longer than 15 seconds with oxygenation as measured per pulse oximetry < 93% and/or transcutaneously measured carbon dioxide partial pressure > 45 mmHg and/ or apnea (defined as cessation of airflow for > 15 seconds)
Number of interventions to regain respiratory stability | Time frame from first applications of intravenous sedatives until finishing the intended procedure
  Number of interventions to reestablish respiratory stability (combined numbers of episode for jaw thrust, repositioning of the patient, repositioning of the patients head, tactile stimulation)
Need for noninvasive ventilation | Time frame from first applications of intravenous sedatives until finishing the intended procedure
  Number of episodes of bag-mask-ventilation
Time of procedure in minutes | Duration of the procedure for which sedation is determined. It covers the time period from first positioning of the patient to repositioning of the patient or patients extremities after completion of the procedure
  Time of procedure in minutes
Time of sedation in minutes | Time frame from first applications of intravenous sedatives until finishing the intended procedure
  Time of sedation in minutes
Use of sedatives | Time frame from first applications of intravenous sedatives until finishing the intended procedure
  Cumulative dose of i.v. sedatives in mg/kg bodyweight/min of procedure
Use of analgesics | Time frame from first applications of intravenous sedatives until finishing the intended procedure
  Cumulative dose of i.v. analgesics in µg/kg bodyweight/min of procedure
Nausea and vomiting | 24 hours after procedural sedation
  Number of Episodes with nausea and/or vomiting within 24 hours after procedural sedation

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Klotz, M.D., Principal Investigator — Center for Pediatrics, Dep. of Pediatric Intensive Care, Medical Center - University of Freiburg, Freiburg, Germany
Locations (1):
- Center for Pediatrics, Pediatric Intensive Care Unit, Procedure Room, Medical Center - University of Freiburg, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deitch K, Chudnofsky CR, Dominici P. The utility of supplemental oxygen during emergency department procedural sedation and analgesia with midazolam and fentanyl: a randomized, controlled trial. Ann Emerg Med. 2007 Jan;49(1):1-8. doi: 10.1016/j.annemergmed.2006.06.013. Epub 2006 Sep 15. PMID 16978741
- [Background] Deitch K, Chudnofsky CR, Dominici P, Latta D, Salamanca Y. The utility of high-flow oxygen during emergency department procedural sedation and analgesia with propofol: a randomized, controlled trial. Ann Emerg Med. 2011 Oct;58(4):360-364.e3. doi: 10.1016/j.annemergmed.2011.05.018. Epub 2011 Jun 15. PMID 21680059